CLINICAL TRIAL: NCT00717938
Title: A Randomized Phase III Study of Standard Treatment +/- Enoxaparin in Small Cell Lung Cancer
Brief Title: A Study of Standard Treatment +/- Enoxaparin in Small Cell Lung Cancer
Acronym: RASTEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number 2007-006033-14
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2016-09

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Cisplatin; Carboplatin; Etoposide; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Standard chemotherapy treatment for patients with small cell lung cancer. Chemotherapy regimen contains a platinum drug and a topoisomerase inhibitor. Numbers of cycles 4-6 according to local variants.Used drugs=cisplatinum or carboplatin and e.g.etoposide.
  Interventions: Drug: cisplatinum or carboplatin and e.g.etoposide.
- B (Experimental): Standard chemotherapy treatment for patients with small cell lung cancer. Chemotherapy regimen contains a platinum drug and a topoisomerase inhibitor. Numbers of cycles 4-6 according to local variants. Used drugs=cisplatinum or carboplatin and e.g.etoposide. In addition to this, subjects will receive daily subcutaneous injections of enoxaparin during chemotherapy treatment.
  Interventions: Drug: cisplatinum or carboplatin and e.g.etoposide+enoxaparin

INTERVENTIONS:
Drug: cisplatinum or carboplatin and e.g.etoposide. — Standard chemotherapy treatment for patients with small cell lung cancer. Chemotherapy regimen contains a platinum drug and a topoisomerase inhibitor. Numbers of cycles 4-6 according to local variants. Used drugs=cisplatinum or carboplatin and e.g.etoposide. Treatment will be given every three weeks for 4-6 cycles according to local variants.
  Other Names: cisplatinum; carboplatin; etoposide
  Arms: A
Drug: cisplatinum or carboplatin and e.g.etoposide+enoxaparin — Standard chemotherapy treatment for patients with small cell lung cancer. Chemotherapy regimen contains a platinum drug and a topoisomerase inhibitor. Numbers of cycles 4-6 according to local variants. In addition to this, subjects will receive daily subcutaneous injections of enoxaparin during chemotherapy treatment.
  Other Names: cisplatinum; carboplatin; etoposide; enoxaparin
  Arms: B

SUMMARY:
The endpoint is to investigate if the addition of low molecular heparin - enoxaparin, will result in a significant increase of overall survival in patients with small cell lung cancer, receiving standard chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy will be given in accordance with local or regional guidelines but shall include a platinum drug + any topoisomerase inhibitor. Within these limits the study will accept different local variants as long as each centre remains consistent to its declared standard chemotherapy regimen. The recommended regimen is carboplatin or cisplatin plus etoposide q3 weeks for 4 cycles but up to 6 cycles is allowed. Local dosages and dose reduction schedules will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically verified SCLC, all stages
2. WHO performance status 0, 1, 2 or 3
3. Age 18 years or older
4. Intention and feasibility to treat with chemotherapy consisting of platinum + topoisomerase inhibitor.
5. Platelets >100 x109 /L
6. Signed informed consent
7. PK (prothrombin complex) INR and APTT within normal ranges.

Exclusion Criteria:

1. Prior systemic chemotherapy for lung cancer.
2. Concomitant anticoagulation treatment, except for ASA or clopidogrel
3. Active overt bleeding of clinical importance or at high risk (e.g. earlier observed haemorrhage in a brain metastasis, severe coagulopathy as haemophilia, severe liver dysfunction with impaired coagulation, acute peptic ulcer, and within the last 3 months suffered from intracranial haemorrhage, or surgery in the central nervous system).
4. Any other known contraindication for enoxaparine ( e.g. Hypersensitivity against enoxaparine and its derivatives).
5. Pregnancy or breast-feeding
6. Fertile women not using effective contraceptives or men who do not agree to use effective contraception during the treatment period.
7. Treatment with any other investigational agent, or participation in any other clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2008-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Significant increase of overall survival | At follow up 1 year after treatment

SECONDARY OUTCOMES:
Toxicity | During treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lars Ek, MD, Principal Investigator — University Hospital, Lund; Jan Sundberg, RN, Study Director — University Hospital, Lund
Locations (16):
- Sweden (16):
  - Gävle hospital, Gävle
  - Sahlgrenska University Hospital, Gothenburg
  - Helsingborg Hospital, Helsingborg
  - Ryhov Hospital, Jönköping, Jönköping
  - Blekinge Hospital, Karlskrona
  - Central Hospital, Karlstad
  - Central Hospital, Kristianstad
  - University Hospital Linköping, Linköping
  - University Hospital Department of Respiratory Medicine, Lund
  - University Hospital MAS, Malmo
  - University Hospital, Örebro, Örebro
  - Karolinska University Hospital, Stockholm
  - Norrlands University Hospital, Umeå
  - Akademiska hospital Uppsala, Uppsala
  - Central Hospital, Vaxjo
  - Ystad hospital, Ystad

REFERENCES:
- [Derived] Ek L, Gezelius E, Bergman B, Bendahl PO, Anderson H, Sundberg J, Wallberg M, Falkmer U, Verma S, Belting M; Swedish Lung Cancer Study Group (SLUSG). Randomized phase III trial of low-molecular-weight heparin enoxaparin in addition to standard treatment in small-cell lung cancer: the RASTEN trial. Ann Oncol. 2018 Feb 1;29(2):398-404. doi: 10.1093/annonc/mdx716. PMID 29106448